CLINICAL TRIAL: NCT00230191
Title: Phase II, Multicenter, Double-Blind, Placebo-Controlled, Parallel-Group, Dose-Ranging Study of the Effects of RK-0202 on Oral Mucositis in Patients Receiving Radiation Therapy for Tumors of the Oral Cavity, Oropharynx, Nasopharynx, Salivary Glands or Supraglottic Region
Brief Title: Safety and Efficacy of RK0202 in Oral Mucositis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RxKinetix (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RK:0202-02; NCT00046956 (obsolete NCT alias)
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Last update posted 2007-01-15 (Estimated); Status verified 2005-10

CONDITIONS: Mouth Diseases; Mouth Ulcers; Oral Mucositis; Head and Neck Cancer
Keywords: Oral; Mucositis; Stomatitis; Head and Neck Cancer
MeSH Terms: conditions — Mouth Diseases; Oral Ulcer; Stomatitis; Head and Neck Neoplasms; Mucositis

INTERVENTIONS:
Drug: RK-0202

SUMMARY:
The primary objective of the study is to assess the effect of RK-0202 versus placebo on the incidence and severity of oral mucositis in subjects receiving radiation therapy for head and neck cancer. Concurrent chemotherapy is not allowed in the study.

DETAILED DESCRIPTION:
Approximately 42,000 new cases of head and neck squamous cell carcinoma occur annually in the United States. Radiotherapy ("RT") plays a significant role in the management of head and neck cancer. The most common and clinically significant toxicities arising from head and neck radiation therapy are acute mucositis and acute and chronic xerostomia (dry mouth or salivary gland changes). In subjects receiving RT for cancers of the oral cavity or oropharynx the incidence of acute mucositis can exceed 90%. The painful ulceration of the oral mucosa produced by the radiation often leads to the requirement for narcotics to control pain, inability to eat, dehydration, the need for parenteral nutrition and, sometimes, breaks in RT. In addition to its symptomatic cost, the presence of mucositis has been associated with a number of other adverse outcomes including higher costs and more frequent hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18 years and older with confirmed tumors of the oral cavity, oropharynx, nasopharynx, salivary glands, or supraglottic region who are intended for treatment with RT alone (no concomitant chemotherapy).
* In post-operative patients, RT must begin no later than 9 weeks following surgery.
* Intended for treatment with an RT regimen that will deliver a minimum of 60 Gy over 5-8 weeks to at least 2cm2 of three or more of seventeen protocol-specific oral cavity anatomical sites. Each qualifying site must receive a minimum of 60 Gy and there must be at least three such sites. (See section 5.3.1). Regimens may consist of:
* single dose daily fractionated (daily max 2.2 Gy)
* hyperfractionated (daily max 2.4 Gy)
* concurrent boost (daily max during boost 3.3 Gy)
* The minimum planned duration of treatment must be 5 weeks and the maximum 8 weeks.
* Ability to undergo oral assessments.
* Ability to begin dosing with study drug on day 1 of RT.
* Karnofsky Performance Score > 60.
* Ability to understand the protocol and provide informed consent.
* If female, have negative serum pregnancy test.

Exclusion Criteria:

* Planned use of concomitant chemotherapy.
* Planned use of amifostine.
* Presence of oral mucositis.
* Prior radiotherapy to the head and neck.
* T1 or T2 glottic tumors.
* Other investigational drugs in the 14 days preceding initiation of study medication or during administration of study medication.
* Other investigational or mucoprotective therapy for the prevention of oral mucositis, including, but not limited to, -carotene, tocopherol, laser irradiation, brushing the oral mucosa with silver-nitrate prophylactically, systemic TGF-β (transforming growth factor beta), misoprostol, pentoxifylline, leucovorin, allopurinol mouthwashes, systemic KGF (keratinocyte growth factor) or pilocarpine. Oral rinses with hydrogen peroxide, sucralfate, or chlorhexidine gluconate are also not permitted during the study.
* Serious recent non-malignant medical condition which, in the opinion of the investigator, makes the patient unsuitable for study participation.
* Medical, sociological, or psychological impediment to probable compliance with protocol.
* Inability to undergo repeat treatments, clinical evaluations and other diagnostic procedures required by the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110
Dates: Start 2003-01; Study Completion 2005-12

PRIMARY OUTCOMES:
The primary objective of the study is to assess the effect of RK-0202 versus placebo on the incidence and severity of oral mucositis.

SECONDARY OUTCOMES:
The secondary objectives of the study are to assess the safety and tolerability of RK-0202 in these subjects and to explore whether the ProGelz™ vehicle alone is active in these subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Sonis, DMD DMSc, Study Director — Harvard, Oral Medicine, Infection & Immunology; Doug Peterson, DMD, Principal Investigator — University of Connecticutt Health Center; Guy Juillard, MD, Principal Investigator — University of California, Los Angeles; Mark Chambers, DMD MS, Principal Investigator — MD Anderson; Andy Trotti, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute; John Feldmeier, DO, Principal Investigator — Medical University of Ohio; Samy El Sayed, MD, Principal Investigator — Ottawa Regional Cancer Centre; Rufus Scrimger, MD, Principal Investigator — Cross Cancer Institute, Edmonton, CA; Jim Wright, MD, Principal Investigator — Juravinski Cancer Centre Hamilton Health Sciences; Donald Welsh, MD, Principal Investigator — Commonwealth ENT, Louisville, KY
Locations (9):
- United States (6):
  - UCLA Medical Center, Los Angeles, California
  - H Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Commonwealth ENT, Louisville, Kentucky
  - University of Connecticutt, Farmington, Massachusetts
  - Medical University of Ohio, Cancer Institute Ruppert Cancer Center, Toledo, Ohio
  - MD Anderson Cancer Center, Houston, Texas
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - Juravinski Cancer Center, Hamilton, Ontario
  - University of Ottawa, Ottawa, Ontario